CLINICAL TRIAL: NCT01890330
Title: Effects of Canola Oil on Vascular and Metabolic Parameters in Individuals With Metabolic Syndrome
Acronym: METCO-2013
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Alberta Innovates Bio Solutions (Other); Alberta Canola Producers Commission (Unknown); Canola Council of Canada (Other)
Responsible Party: Principal Investigator, Dr. Carla Taylor, Professor and Principal Investigator, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: B2013:006
Record Dates: First submitted 2013-06-03; First posted 2013-07-01 (Estimated); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Metabolic Syndrome
Keywords: Canola Oil; Metabolic Syndrome; Serum LDL cholesterol
MeSH Terms: conditions — Metabolic Syndrome | interventions — Rapeseed Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Canola Oil 25 g/d (Experimental): Participants randomized to this arm will be provided with food items including entrées, side dishes, salad dressing, baked goods, and desserts prepared with traditional canola oil to incorporate into their usual eating pattern. They will consume one or two food items per day containing a total of 25 g/d of Canola oil.
  Interventions: Other: Canola Oil 25 g/d
- Non-Canola Oil Mixture 25 g/d (Active Comparator): Participants randomized to this arm will be provided with food items including entrées, side dishes, salad dressing, baked goods, and desserts prepared with an oil mixture representing the typical Western diet to incorporate into their usual eating pattern. They will consume one or two food items per day containing a total of 25 g/d of the non-canola oil mixture.
  Interventions: Other: Non-Canola Oil Mixture 25 g/d

INTERVENTIONS:
Other: Canola Oil 25 g/d — Daily consumption of food items containing traditional canola oil (25 g/d) for 12 weeks.
  Arms: Canola Oil 25 g/d
Other: Non-Canola Oil Mixture 25 g/d — Daily consumption of food items containing Non-Canola Oil Mixture (25 g/d) representing the typical Western diet for 12 weeks.
  Arms: Non-Canola Oil Mixture 25 g/d

SUMMARY:
MetS is an early stage of CVD and is an appropriate target for dietary interventions. MetS is a clustering of risk factors (abdominal obesity, elevated serum triglycerides, low HDL-cholesterol, hypertension, elevated fasting blood glucose) accompanied by low grade chronic inflammation, hepatic steatosis (fatty liver) and reduced vascular function.

This study will investigate the effect of a 12 week intervention with canola oil versus the typical fat mixture in the Western diet on blood lipids, blood vessel function and MetS parameters. CVD risk will be assessed based on the profile of lipids and other factors in the blood as well using specialized equipment for non-invasive monitoring of blood vessel function.

DETAILED DESCRIPTION:
The current, worldwide obesity epidemic is significantly increasing the number of individuals with Metabolic Syndrome (MetS), an early stage combination of risk factors which predisposes individuals to cardiovascular disease (CVD) and other chronic diseases. While it has been shown that modification of dietary fat intake can play an important role in prevention and management of CVD there is an absence of dietary intervention studies focusing on dietary oils and early stage modification of MetS components, particularly those affecting progression to CVD.

The composition of canola oil is considered healthy. However, there is a lack of scientifically sound clinical studies directly comparing canola oil with other fats in the diet. Given that much of the evidence for current dietary recommendations for type and amounts of fatty acids is based on heart disease, the proposed research will contribute to the knowledge base for dietary fat recommendations for individuals with MetS.

Specifically, this study will investigate the effect of a 12 week intervention with canola oil versus the typical fat mixture in the Western diet on blood lipids, blood vessel function and MetS parameters. CVD risk will be assessed based on the profile of lipids and other factors in the blood as well using specialized equipment for non-invasive monitoring of blood vessel function.

ELIGIBILITY:
Inclusion Criteria:

1. Male, or non-pregnant, non-lactating females, aged 20 - 75 years;
2. LDL-Cholesterol >2.5 mmol/L and <5.0 mmol/L
3. If the participant has 2 or more of the following characteristics of MetS

   * Fasting blood glucose >5.6 mmol/L and <7.0 mmol/L;
   * Blood pressure >130/85 mm Hg and <150/100;
   * Triglycerides >1.7 mmol/L and <4.0 mmol/L;
   * HDL-cholesterol <1.0 mmol/L in males or <1.3 mmol/L in females;
   * Abdominal obesity as defined by a waist circumference of >102 cm (40 inches) in males and >88 cm (35 inches) in females of non-Asian ethnicity, and a waist circumference of >94 cm (37 inches) in males and >80 cm (32 inches) in females of Asian ethnicity.
4. Able to read, write and communicate orally in English;
5. Willing to maintain a stable level of activity during participation in the study;
6. Willing to maintain dietary routine, refrain from consuming omega-3 supplements or omega-3 rich foods (>0.3 grams ALA/serving or, >0.1 grams of EPA and DHA; see handout with examples) and refrain from taking any over-the-counter medications or herbal supplements specified for weight loss, or the lowering of blood lipids, blood glucose or blood pressure from acceptance into the study until the final study visit;
7. Willing to comply with protocol requirements and procedures;
8. Willing to provide written informed consent.

Exclusion Criteria:

1. Use of prescribed medications for lowering or managing blood lipids (hyperlipidemia), blood glucose (hyper/hypoglycemia), blood pressure (hypertension) or body weight;
2. Regular use of non-prescription products, over-the-counter medications, or herbal supplements designed to lower blood lipids, blood glucose, blood pressure or body weight, or omega-3 supplements or omega-3 rich foods, within the past 3 months;
3. Participating in or adhering to a weight loss diet or physical activity program designed to facilitate weight loss.
4. Adhering to a physician or dietitian directed lifestyle or dietary modification program for the purpose of lowering hypercholesterolemia;
5. Medical history of liver disease, with the exception of fatty liver, or chronic renal disease;

5. Any acute medical condition or surgical intervention within the past 3 months; 6. Conditions or medications which are likely to increase the risk to the participants or study personnel, or to reduce the ability of the participant to comply with the protocol, or affect the results; 7. History of gastrointestinal reactions or allergies to canola oil or to one or more ingredients in the study foods which significantly limits the number of study foods that can be consumed; and 8. Currently participating in or having participated in a food intervention study within the last 3 months.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in Fasting Serum LDL-cholesterol | Baseline, Week 6 and Week 12
  Fasting blood sample will be taken at Baseline (Day 1), Week 6 (Day 56) amd Week 12 (Day 84) for purpose of analysis of Serum LDL-Cholesterol.

SECONDARY OUTCOMES:
Change in Blood Vessel Function | Baseline, Week 6 and Week 12
  Blood vessel function will assessed and compared at Baseline (Day 1), Week 6 (Day 56) and Week 12 (Day 84) via pulse wave analysis and pulse ave velocity.
Change in Total Cholesterol | Baseline, Week 6, and Week 12
  A fasting blood sample will be obtained at Baseline (Day 1), Week 6 (Day 56) and Week 12 (Day 84) for analysis and comparison of serum total cholesterol
Change in Advanced Glycation Endproducts (AGEs) | Baseline, Week 6, and Week 12
  Advanced Glycation Endproducts (AGEs) will be obtained and compared at Baseline (Day 1), Week 6 (Day 56), and Week 12 (Day 84) using the AGE Reader.
Change in Biomarkers of Vascular Function | Baseline, Week 6 and Week 12
  A fasting blood sample will be obtained at Baseline (Day 1), Week 6 (Day 56), and Week 12 (Day 84) for the assessment and comparison of biomarkers of vascular function, inflammation, oxidative stress, and immune function.
Change in Total Body Fat Composition | Baseline and Week 12
  Participants will undergo a body composition scan using a GE Lunar Dual Energy X-Ray Absorptiometry scanner to determine the percentage of total body fat, abdominal fat, and percentage of lean muscle mass at Baseline (Day 1) and Week 12 (Day 84).
Change in Fatty Liver | Baseline and Week 12
  Fatty liver will be assessed through serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST).
Change in Anthropometrics | Baseline, Week 6 and Week 12
  Weight, body mass index (BMI), and waist circumference and will be obtained and compared at with Baseline (Day 1), Week 6 (Day 56) and Week 12 (Day 84).
Change in HDL-Cholesterol | Baseline, Week 6, and Week 12
  A fasting blood sample will be obtained at Baseline (Day 1), Week 6 (Day 56) and Week 12 (Day 84) for analysis and comparison of HDL-cholesterol.
Change in Triglycerides | Baseline, Week 6, and Week 12
  A fasting blood sample will be obtained at Baseline (Day 1), Week 6 (Day 56) and Week 12 (Day 84) for analysis and comparison of serum triglycerides.
Change in Fasting Blood Glucose | Baseline, Week 6 and Week 12
  A fasting blood sample will be obtained at Baseline (Day 1), Week 6 (Day 56) and Week 12 (Day 84) for analysis and comparison of glucose.
Change in Fasting Insulin | Baseline, Week 6 and Week 12
  A fasting blood sample will be obtained at Baseline (Day 1), Week 6 (Day 56) and Week 12 (Day 84) for analysis and comparison of insulin (and calculation of insulin sensitivity using HOMA-IR, QUICKI).
Change in Glycated Hemoglobin (HbA1c) | Baseline, Week 6 and Week 12
  A fasting blood sample will be obtained at Baseline (Day 1), Week 6 (Day 56) and Week 12 (Day 84) for analysis and comparison of glycated hemoglobin (HbA1c).
Change in fasting C-reactive protein | Baseline, Week 6 and Week 12
  A fasting blood sample will be obtained at Baseline (Day 1), Week 6 (Day 56) and Week 12 (Day 84) for analysis and comparison of C-reactive protein.

CONTACTS AND LOCATIONS:
Overall Officials: Carla Taylor, PhD, Principal Investigator — University of Manitoba
Locations (1):
- St. Boniface General Hospital - I.H. Asper Clinical Research Institute, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Despres JP, Lemieux I. Abdominal obesity and metabolic syndrome. Nature. 2006 Dec 14;444(7121):881-7. doi: 10.1038/nature05488. PMID 17167477
- [Result] Jakobsen MU, O'Reilly EJ, Heitmann BL, Pereira MA, Balter K, Fraser GE, Goldbourt U, Hallmans G, Knekt P, Liu S, Pietinen P, Spiegelman D, Stevens J, Virtamo J, Willett WC, Ascherio A. Major types of dietary fat and risk of coronary heart disease: a pooled analysis of 11 cohort studies. Am J Clin Nutr. 2009 May;89(5):1425-32. doi: 10.3945/ajcn.2008.27124. Epub 2009 Feb 11. PMID 19211817
- [Derived] Pauls SD, Du Y, Clair L, Winter T, Aukema HM, Taylor CG, Zahradka P. Impact of Age, Menopause, and Obesity on Oxylipins Linked to Vascular Health. Arterioscler Thromb Vasc Biol. 2021 Feb;41(2):883-897. doi: 10.1161/ATVBAHA.120.315133. Epub 2020 Dec 31. PMID 33380172
- See also: Canadian Centre for Agri-Food Research in Health and Medicine — http://www.ccarm.ca